CLINICAL TRIAL: NCT01321229
Title: Influence of the Sleep Apnea Syndrome on the Functional Recovery After Stroke in a Rehabilitation Unit
Brief Title: The Influence of the Sleep Apnea on the Neurological and Functional Recovery
Acronym: SAS-AVC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: UC0902
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2012-11

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep apnea; NIHSS scale; FIM scale; FUGL-MEYER scale
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With sleep APNEA: Sleeping Apnea Syndrome (SAS) screening usin an APNEA LINK device within the 10 first days following the admission Diagnosis and medical care by a sleeping disorder qualified specialist
- Without sleep APNEA: Sleeping Apnea Syndrome (SAS) screening usin an APNEA LINK device within the 10 first days following the admission

SUMMARY:
The sleep respiratory troubles (central apnea or CHEYNES-Stokes dyspnea) are frequent after stroke. The association of the sleep respiratory troubles with a reserved functional prognosis is debated. The purpose is to find out the frequency of the sleep respiratory troubles after stroke in a PRM department and to study their relationship with functional and neurological recovery.

DETAILED DESCRIPTION:
The sleep respiratory troubles (central apnea or CHEYNES-Stokes dyspnea) are frequent after stroke. The association of the sleep respiratory troubles with a reserved functional prognosis is debated. The purpose is to find out the frequency of the sleep respiratory troubles after stroke in a PRM department and to study their relationship with functional and neurological recovery.

Forty-five patients with the average of 58,2 years had been included in this prospective MONOCENTRICAL study. The detection of the sleep respiratory troubles was realised using a nocturnal oxymetry device and measuring the inspiratory flow, gathering the index of apnea-hypopnea.

The NIHSS, the FIM and the FUGL-MEYER scales were used at the moment of inclusion and two months AFTERWORDS.

ELIGIBILITY:
Inclusion Criteria:

Patient's or one family member's agreement for participation in the study Being aged over 18 years Stroke history in the past 6 months (ischemic or hemorrhagic) Hospitalisation in PRM department and participation to a rehabilitation program during study Patient belonging to the social security system

Exclusion Criteria:

Patient having a sleep apnea syndrome known prior to inclusion Patient presenting a cardiorespiratory INSUFIENCY Patients being INABLE to carry-out the tests or presenting a mental disorder Patients who started already their rehabilitation program before in another PRM center or department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke history in the past 6 months (ischemic or hemorrhagic) and Hospitalisation in PRM department and participation to a rehabilitation program during study
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
the variation of the FIM (Functional Independence Measure) | at 2 months
  defined by the FIM score after 2 months minus the FIM score at the initial moment(T0)

SECONDARY OUTCOMES:
age | at inclusion
BMI (Body Mass Index) | at inclusion
Score NIHSS (National Institute of Health Stroke Score) | at 2 months
  Comparison between inclusion and 2 months
Fugl Meyer Assessment of Motor Recovery after Stroke | at 2 months
  comparison between inclusion and 2 months
Epworth Sleepiness Scale (ESS) | at inclusion
Attention tests | at inclusion
  BAWL Test (Batterie Attentionnelle William Lennox)

CONTACTS AND LOCATIONS:
Overall Officials: Alain YELNIK, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- PRM Department, Hôpital Fernand Widal - Pr Alain YELNIK, Paris, France